CLINICAL TRIAL: NCT05898997
Title: Regulation of Intraocular Pressure in Glaucoma Patients by Acupressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202303119RINA
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-04

CONDITIONS: Primary Open Angle Glaucoma; Acupressure
Keywords: Primary Open Angle Glaucoma; High intraocular pressure; Acupressure; Bladder Meridian; Triple Burner Meridian
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: The patients included in the study were between the ages of 15 and 80 and were classified into 5 groups based on their visual field defect levels.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Normal (Visual Field Defects: >-2.00 dB) (Experimental): Do the formal acupressure
  Interventions: Behavioral: Acupressure
- Mild (Visual Field Defects: -2.00~-6.00 dB) (Experimental): Do the formal acupressure
  Interventions: Behavioral: Acupressure
- Moderate (Visual Field Defects: -6.01~-12.00 dB) (Experimental): Do the formal acupressure
  Interventions: Behavioral: Acupressure
- Severe (Visual Field Defects: -12.01~-20.00dB) (Experimental): Do the formal acupressure
  Interventions: Behavioral: Acupressure
- Profound (Visual Field Defects: <-20 dB) (Experimental): Do the formal acupressure
  Interventions: Behavioral: Acupressure

INTERVENTIONS:
Behavioral: Acupressure — Massage the following acupoints in order: Jing Ming, Zan Zhu, Mei Chong, Yu Yao, and Si Zhu Kong. Use the joint of your thumb to massage each acupoint for 30 times, and repeat the cycle at least once. Then, continue to promote the circulation of qi by gently making a fist and using the four fingers to scrape along the upper eye socket from inside to outside. Scrape each side 30 times, and do it separately for the left and right sides. It is recommended to do this process at least once in the morning and once in the evening.
  Other Names: Acupuncture point massage

SUMMARY:
The purpose of this clinical trial is to implement acupressure twice daily and monitor the changes in intraocular pressure (IOP) in patients with different levels of glaucoma. The study aims to investigate the effects of this method on IOP, visual field, retinal nerve fiber layer thickness measured by optical coherence tomography, blood vessel density, and macular ganglion cell layer thickness and density in patients with primary open-angle glaucoma (POAG).

DETAILED DESCRIPTION:
[Background] With the advancement of medical technology, many diseases can be controlled through Western medicine. However, there are still some diseases that cannot be effectively treated with Western medicine alone. Therefore, this article approaches the treatment of glaucoma from the perspective of traditional Chinese medicine meridians, by using acupressure to verify its effectiveness in reducing intraocular pressure in glaucoma patients.

[Participants] Between May 2023 and February 2024, a total of 80 patients were randomly selected from the ophthalmology outpatient clinic of National Taiwan University Hospital Hsinchu Branch. The patients included in the study were between the ages of 15 and 80 and were classified into 5 groups based on their intraocular pressure (IOP) levels.

The inclusion criteria were primary open-angle glaucoma and high IOP. Patients with angle-closure glaucoma, and those who had previously undergone eye surgery were excluded from the study.

[Materials and Methods] Massage the following acupoints in order: Jing Ming, Zan Zhu, Mei Chong, Yu Yao, and Si Zhu Kong. Use the joint of your thumb to massage each acupoint for 30 times, and repeat the cycle at least once. Then, continue to promote the circulation of qi by gently making a fist and using the four fingers to scrape along the upper eye socket from inside to outside. Scrape each side 30 times, and do it separately for the left and right sides. It is recommended to do this process at least once in the morning and once in the evening.

[Postoperative follow-up and evaluation] After one week, the best corrected visual acuity and changes in intraocular pressure will be followed up, and changes in intraocular pressure will be monitored regularly at 1 month, 3 months, 6 months, 9 months, and 12 months. Visual field testing and optical coherence tomography (OCT) will be monitored regularly at 6 months and 12 months.

[Data Statistics and Analysis] Record the subjects' intraocular pressure and visual acuity for statistical analysis. IBM SPSS v21.0 statistical software (IBM Corporation, New York, USA) will be used to calculate descriptive statistics, including mean ± standard deviation (±SD), median, range, and frequency and percentage as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary open-angle glaucoma, normal-tension glaucoma, and high intraocular pressure.

Exclusion Criteria:

* Patients with narrow-angle glaucoma, patients who have undergone eye surgery during the study period, patients who are unable to learn the acupoint massage procedure or unable to perform it regularly.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure changes | Monitored regularly at 1 week, 1 month, 3 months, 6 months, 9 months, and 12 months.
  Tracking the intraocular pressure changes in patients with different stages of glaucoma after undergoing acupoint massage

SECONDARY OUTCOMES:
Visual field testing by optical coherence tomography (OCT) | Monitored at 6 months and 12 months.
  Tracking the changes of visual field testing by optical coherence tomography (OCT) in patients with different stages of glaucoma after undergoing acupoint massage

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No
Undecided